CLINICAL TRIAL: NCT06431711
Title: Fundus Optical coheRence Tomography Angiography Evaluation for Small-vessel Health in Cerebral Small Vessel Disease
Acronym: FRESH-CSVD
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024050
Record Dates: First submitted 2024-04-25; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Small Vessel Diseases; Retinal Ischemia; Choroid; Injury
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with CSVD: This does not entail the application of interventions.

SUMMARY:
Cerebral small-vessel disease (CSVD) is a significant contributor to stroke and dementia, primarily impacting individuals over the age of 60. Its prevalence exceeds 70% in the elderly population, imposing a substantial burden on brain health and the economy. Optical coherence tomography angiography (OCTA) is a new type of optical diagnostic imaging technology for non-invasive detection, which can perform multi-dimensional quantitative assessment of fundus retinopathy. Current studies have shown that fundus OCTA-derived parameters may have potential in characterizing imaging changes in CSVD. However, the correlation between retinal/choroidal parameters on OCTA and the CSVD imaging markers remains uncertain. FRESH-CSVD is a prospective, observational study that will use fundus OCTA-derived parameters to screen patients with CSVD, explore the relationship between relevant parameters based on OCTA measurements and CSVD, and evaluate the feasibility and clinical value of identification of CSVD through fundus OCTA.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 35 years old;
2. Patients who underwent Multimodal MRI with any CSVD imaging marker;
3. Subjects who have signed informed consent.

Exclusion Criteria:

1. Patient who was unable to cooperate with examinations;
2. There are known diseases that may cause or worsen CSVD (brain injury, Down syndrome, Alzheimer's disease, Parkinson's disease, etc.);
3. There are known eye diseases or severe underlying fundus lesions that may impact fundus assessment;
4. Suffering from serious systemic diseases, such as heart, liver, kidney diseases or major mental illnesses;
5. Contraindications for imaging examinations

Exit Criteria:

1. Not meet the inclusion criteria.
2. For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator.
3. Any adverse or serious adverse events during the study period judged by investigator

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research population for this study consists of patients who have been diagnosed with non-acute ischemic symptoms of Cerebral Small Vessel Disease. Inclusion criteria: Patients with any of the CSVD-related MRI imaging markers; Patients aged old than 35 years; Sign informed consent. Exclusion criteria: Unable to cooperate with examinations; Known dementia; Serious systemic illness; Contraindications for imaging examination; Known retinal diseases. Exit criteria: not meet the inclusion criteria; For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator; Any adverse or serious adverse events during the study period judged by investigator.
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2034-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of fundus OCTA-derived parameters for CSVD | baseline ,6-month, and every 1 year, follow-up time up to 5 years
  Investigators intend to use these indicators to assess the diagnostic accuracy of fundus OCTA for CSVD: area under the receiver operating characteristic curve (AUROC)

SECONDARY OUTCOMES:
The development of total CSVD burden in MRI | baseline ,6-month, and every 1 year, follow-up time up to 5 years
  Total brain small-vessel disease burden is used to assess the overall impact of CSVD, with a score range of 0-4 points
Number of Patients with cerebrovascular events, cardiovascular events, dementia or death | baseline ,6-month, and every 1 year, follow-up time up to 5 years
  Cerebrovascular events included ischemic stroke, transient ischemic attack (TIA) and cerebral hemorrhage. Cardiovascular events included angina and myocardial infarction.
  Using the Chinese version of the MMSE scale, dementia is defined based on different levels of education (≤ 22, ≤ 23, ≤ 24, ≤ 26 points for illiteracy, primary school, junior high school, and university).
  Death included any reason caused death.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No